CLINICAL TRIAL: NCT01375621
Title: Epidemiology of Rural MRSA : Is Livestock Contact a Risk Factor?
Brief Title: Livestock Contact and MRSA in Rural Areas
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911169; 11-C-N169
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Staphylococcus Aureus Infection
Keywords: Farming; Antibiotic Resistant; Bacteria
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- AHS cohort: population of S. aureus asymptomatic rural Iowans
- Non-AHS group: symptomatic S. aureus infections in rural Iowans.

SUMMARY:
Background:

- MRSA is a type of bacteria that causes serious health problems. It can cause severe infections and is difficult to treat. MRSA has been found in a high number of people who work with some kinds of livestock, such as pigs. Researchers want to study people in rural areas, where more people work with or around livestock. They want to see if MRSA is more common or causes more serious infections in these areas.

Objectives:

- To look at the relationship between livestock handling (especially pigs) and MRSA bacteria in people in rural areas.

Eligibility:

* Participants in the Agricultural Health Study in Iowa, including those who are exposed to livestock.
* Healthy volunteers who are not exposed to livestock.

Design:

* This study requires an initial visit and monthly follow-up surveys for 18 months.
* At the first visit, participants will have throat and nose swabs to collect cell and bacteria samples. They will also complete a questionnaire about their health habits. Other questions will ask about any work that brings them into contact with livestock like cows, pigs, or chickens.
* Every month for the next 17 months, participants will complete another questionnaire to record any changes in their health and livestock contact information. They will also collect throat and nose swabs. They will send the questionnaires and the swabs to the study researchers.
* Participants will be paid for the first visit and for every monthly survey and swab collection they return.
* No treatment will be given as part of this protocol.

DETAILED DESCRIPTION:
The goal of this study is to understand the epidemiology of antibiotic-resistant S. aureus, including methicillin resistant S. aureus (MRSA), outside of the hospital environment. Our objective is to characterize the epidemiology of S. aureus in the rural community, focusing on persons who have contact with livestock. We will achieve this by carrying out two parallel prospective cohort studies in Iowa, examining 1) individuals enrolled in the Agricultural Health Study, including those who raise swine; and 2) a matched population-based group with no livestock exposure. We will partner with the state s microbiological diagnostic laboratories in order to collect isolates from the symptomatic S. aureus infections. Our central hypothesis is that individuals working in close proximity to livestock and poultry are at risk of occupational exposure to MRSA. We further hypothesize that farmers in contact with livestock (swine in particular) will be more likely to be colonized with swine-associated S. aureus strains than are individuals without contact. Finally, we expect to see both typical human strains of S. aureus (including USA300) as well as animal-associated strains (such as ST398) causing infections in Iowans. Our rationale is that successful completion will provide opportunities to institute an early warning system to evaluate emerging S. aureus strains, allowing for potential interventions prior to widespread dissemination in the human population. We will test our central hypothesis and accomplish the objective of this application by pursuing the following specific aims:

1. Establish the prevalence, molecular subtypes, and antibiotic resistance profiles of S. aureus in populations of rural Iowans, and determine risk factors for colonization. We hypothesize that individuals in contact with swine will be more likely to carry MRSA than individuals lacking such exposure; that swine workers will more frequently be colonized with swine-associated strains such as ST398; and that S. aureus isolates collected from livestock farmers will more frequently demonstrate resistance to antibiotics including methicillin and tetracyclines than isolates collected from individuals lacking livestock exposure.
2. Determine the incidence and molecular epidemiology of symptomatic S. aureus infections in rural Iowans. We hypothesize that symptomatic infections will be uncommon in our cohort relative to colonization, and that the majority of such infections will be skin and soft tissue infections. We further hypothesize that the majority of infections in our cohorts and elsewhere in the state will be caused by common strains (including USA300), but that some infections will also be caused by animal-associated strains, including ST398.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Cohort A: Participant or child of participant in the Agricultural Health Study
* Cohort B: Resident of Iowa

EXCLUSION CRITERIA:

* Cohort A: Age <8 months
* Cohort B: Age <8 months

Ages: 6 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals enrolled in the Agricultural Health Study, including those who raise swine; and a matched population-based group with no livestock exposure.
Sampling Method: Non-Probability Sample
Enrollment: 1342 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Epidemiology of MRSA in AHS cohort | ongoing
  Establish the prevalence, molecular subtypes, and antibiotic resistance profiles of S. aureus in populations of rural Iowans, and determine risk factors for colonization.
Epidemiology of MRSA in matched, population-based non-AHS group | ongoing
  Determine the incidence and molecular epidemiology of symptomatic S. aureus infections in rural Iowans.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Beane-Freeman, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Iowa, Coralville, Iowa, United States

REFERENCES:
- [Background] Graham PL 3rd, Lin SX, Larson EL. A U.S. population-based survey of Staphylococcus aureus colonization. Ann Intern Med. 2006 Mar 7;144(5):318-25. doi: 10.7326/0003-4819-144-5-200603070-00006. PMID 16520472
- [Background] Wertheim HF, Melles DC, Vos MC, van Leeuwen W, van Belkum A, Verbrugh HA, Nouwen JL. The role of nasal carriage in Staphylococcus aureus infections. Lancet Infect Dis. 2005 Dec;5(12):751-62. doi: 10.1016/S1473-3099(05)70295-4. PMID 16310147
- [Background] Fritz SA, Epplin EK, Garbutt J, Storch GA. Skin infection in children colonized with community-associated methicillin-resistant Staphylococcus aureus. J Infect. 2009 Dec;59(6):394-401. doi: 10.1016/j.jinf.2009.09.001. Epub 2009 Sep 9. PMID 19747505